CLINICAL TRIAL: NCT01135732
Title: Cytological Evaluation of Biliary Epithelium After Previous Endoscopic Sphincterotomy for Benign Disease
Brief Title: Cytological Evaluation of Biliary Epithelium After Endoscopic Sphincterotomy
Status: Completed | Type: Observational
Sponsor: University of Athens (Other)
Responsible Party: John Kalaitzis MD, Tzaneio General Hospital
Other Study IDs: 10438
Record Dates: First submitted 2010-06-01; First posted 2010-06-03 (Estimated); Last update posted 2010-11-16 (Estimated); Status verified 2009-10

CONDITIONS: Endoscopic Sphincterotomy; Cholangiocarcinoma
Keywords: late development cholangiocarcinoma
MeSH Terms: conditions — Cholangiocarcinoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- study group-previous sphincterotomy
  Interventions: Procedure: brush cytology
- control group-not previous sphincterotomy
  Interventions: Procedure: brush cytology

INTERVENTIONS:
Procedure: brush cytology — brush cytology during ERCP

SUMMARY:
PROTOCOL

Introduction: The introduction of endoscopic retrograde cholangio-pancreatography (ERCP) and endoscopic sphincterotomy (ES) in 1974 has dramatically changed the treatment of biliary and pancreatic diseases. ES permits transection of Oddi's sphincter, allowing the endoscopist to remove stones and place stents.

The main indications for ERCP are: 1. Removal of common bile duct stones 2. Dilation of benign biliary ducts strictures 3. Stent placement in patients with malignancy 4. Acute biliary pancreatitis 5. Removal of stones and dilation of strictures of the main pancreatic duct in patients with chronic pancreatitis and 6. Treatment of biliary fistulae after surgical operations .

Complications of ES can be described as early (within one month after ES) and late. Early complications have approximately a 10% incidence and include: 1.acute pancreatitis (5,4%) 2.bleeding (2%) 3.acute cholangitis (1%) 4.acute cholecystitis (0,5%) 5. Perforation and others (1,1%). Late complications are mainly the recurrence of choledocholithiasis (2,5%), narrowing of the previous ES and recurrent acute cholangitis. Furthermore, there is a debate in the literature about late development of cholangiocarcinoma.

Carcinogenesis after surgical sphincteroplasty and biliary-enteric anastomosis has been described. Previous studies have shown late development of cholangiocarcinoma after transduodenal sphincteroplasty and biliary-enteric anastomosis for benign disease. The incidence is up to 7% in a twenty-year follow up, while in the general population is approximately 1/ 100.000 . In addition, Tocchi et al showed that the rate of cholangiocarcinoma after transduodenal sphincteroplasty and choledochoduodenal anastomosis is up to 5-7% and after other choledochi-enteric anastomoses approximately 1,9%. It seems that the ablation of sphincter function causes prolonged pancreatobiliary and duodenobiliary reflux. Proteolytic pancreatic enzymes are activated and bacterial intestinal flora colonizes the biliary epithelium, causing recurrent inflammation. Chronic inflammatory irritation may lead to hyperplasia, dysplasia and atypia of epithelium, ultimately inducing carcinogenesis.

Eleftheriadis et al, studied changes of the biliary epithelium in patients who underwent choledochi-duodenal anastomosis for benign disease, and hyperplasia of the biliary epithelium was demonstrated. The same results and atypia of biliary epithelium were reported by Kurumado et al, in mice models with choledochi-duodenal anastomosis. Anomalous pancreatobiliary junction and choledochal cysts produce the same histologic alterations of the biliary epithelium.

These facts raise a great amount of concern about late development of cancer after ES. Bergman et al in a small trial argues that after ES, the function of the biliary sphincter is permanently lost. On the other hand, Sugiyama et al demonstrated the reduction of pancreatobiliary reflux 1 year after ES. In addition, large population-based studies have shown no causal association between ES and cholangiocarcinoma, but with enough limitations in study design. In conclusion, the long term cytologic changes of the biliary epithelium after ES for benign disease are not well known.

During ERCP, brush cytology can be performed to evaluate bile duct strictures. The use of endoscopic brushing after ES has no reported complications .

Objective: To evaluate cytologic alterations of the biliary epithelium after previous endoscopic sphincterotomy for benign disease.

DETAILED DESCRIPTION:
Informed consent will be obtained from all patients. ERCP will be conducted at the Endoscopic Unit of Aretaieion University Hospital and Tzaneio General Hospital, Athens, Greece. Pethidine, midazolam or propofol will be used for patient sedation. ERCP will be conducted with the use of a side viewing endoscope. After catheterization of the common bile duct through the previous sphincterotomy, cellular material will be obtained with the use of an endoscopic brush from the bile ducts. With the same way, brush cytology will be performed in the control group after performing ES.

Material obtained from each patient will be smeared on five glass slides. Four slides will be fixed with ethanol solution 95% and the fifth will be air dried. The brush will be fixed in suitable liquid for performing liquid phase cytology. Immunocytology with immunofluorescence p-53 antibody will be performed in samples with hyperplasia, dysplasia or atypia. The cytology department of Tzaneio Hospital will conduct examination and evaluation of all samples.

Samples based on their morphological characteristics will be classified in five categories: a. inadequate sample (very small cell number, presence of blood, inadequate fixation) b. negative for malignancy (adequate cell number with benign morphologic characteristics) c. reactive with or without atypia (cells with reactive/proliferative or inflammatory characteristics. Malignancy is rare but cannot be excluded) d. suspicious for malignancy e. positive for malignancy [21,22].

Examination and evaluation of the specimens will be done by two specialized cytologists, separately, in order to achieve more objective results.

ELIGIBILITY:
inclusion criteria

* age >18
* perform endoscopic sphincterotomy
* benign disease
* cholelithiasis
* biliary colic
* choledocholithiasis
* cholangitis
* biliary pancreatitis

exclusion criteria

* biliary stricture
* malignancy any kind

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients undergoing ERCP and ES for benign disease
Sampling Method: Non-Probability Sample
Enrollment: 56 (Estimated)
Dates: Start 2006-10; Primary Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Athens Medical School, Athens, Greece